CLINICAL TRIAL: NCT01821950
Title: Evaluation of Yoga for Substance Use Risk Factors in a School Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Kripalu Center for Yoga and Health (Other); Boston University (Other)
Responsible Party: Principal Investigator, Sat Bir Khalsa, PhD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007P002600B; R34DA032756 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Adolescent Development
Keywords: Mental health; Substance use; Substance use initiation; Education; Mind Body Therapies; Yoga; Meditation; Adolescent; Adolescence; Child; Children; Middle School
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical education as usual (No Intervention): Physical education curriculum established by the school, including competitive sports, aerobic and anaerobic activities, balance and coordination skills. Yoga is not a component of the curriculum.
- Yoga during physical education (Experimental): 12 to 16 weeks of group yoga classes (approximately 32 classes per student), 30-45 minutes per class, 2-3 times per week, during physical education class. Yoga program includes physical postures and movement, breathing exercises, partner/group games, deep relaxation and meditative techniques.
  Interventions: Behavioral: Yoga during physical education

INTERVENTIONS:
Behavioral: Yoga during physical education — 12 to 16 weeks of group yoga classes (approximately 32 classes per student), 30-45 minutes per class, 2-3 times per week, during physical education class. Yoga program includes physical postures and movement, breathing exercises, partner/group games, deep relaxation and meditative techniques.
  Other Names: Kripalu Yoga In The Schools
  Arms: Yoga during physical education

SUMMARY:
This study will evaluate the efficacy of yoga taught during school to positively influence risk and protective factors of substance use and the initiation and severity of substance use. The study hypothesis is that, compared to a control group participating in regular physical education classes, subjects who participate in 32 yoga sessions across an academic year will improve in negative internalizing behaviors and self-regulatory skills that are known risk and protective factors for substance use. This study will also test the hypothesis that the yoga intervention will reduce both severity of substance use and the degree of substance use initiation.

DETAILED DESCRIPTION:
The long-term, programmatic goal of this research is to advance prevention of addictive behaviors especially substance use in normal adolescent psychological development. The overall goal of this proposal is to pilot test a novel, preventive intervention for adolescent substance use. More specifically, it will evaluate the efficacy of yoga taught during school to positively influence risk and protective factors of substance use and the initiation and severity of substance use.

This study involves a group randomized, controlled trial of yoga compared to physical education-as-usual for one school year, with a 6-month and 1-year follow-up, in order to accomplish the following specific aims:

Specific Aim 1 - To evaluate the efficacy of a school-based yoga program for reducing negative internalizing behaviors (negative mood, perceived stress, impulsivity) which are risk factors for adolescent substance use.

Specific Aim 2 - To evaluate the efficacy of this yoga program for promoting self-regulatory skills as protective factors against substance use in adolescence.

Specific Aim 3 - To conduct a preliminary evaluation of the efficacy of this yoga program for reducing substance use initiation and severity of use.

ELIGIBILITY:
Inclusion Criteria:

* Registered for physical education class

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in self-reported mood as measured by the 24-item Brunel University Mood Scale (BRUMS, total and 6 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  The Brunel University Mood Scale (BRUMS) will be used to measure change in self-reported mood. The BRUMS is designed specifically for assessing mood in adolescents. It contains 24 adjectives that are all rated on a four-point scale to give a total mood score and scores for six subscales: tension, depression, anger, vigor, fatigue, and confusion. In a validation sample of nearly 2,000 British adolescents (12 to 18 years of age), multi-sample confirmatory factor analysis showed high factor validity. Criterion and construct validity were also acceptable. Furthermore, BRUMS is sensitive to short-term changes. More recently, the BRUMS has been successfully used in a large sample of American adolescents. Negative affective states, such as mood, are clearly linked to substance use trajectories.
Change in self-reported stress levels as measured by the 10-item Perceived Stress Scale (PSS) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the degree to which events are appraised as stressful during the last month. Construct and convergent validity is adequate, since it is moderately correlated with other measures of stress and self-reported health status. The 10 items in this scale were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. It is psychometrically sound based on epidemiological sampling that evaluated reliability and validity. Furthermore, the PSS has been administered to mid-adolescents (8th and 9th graders) with good internal consistency. Psychological stress has been associated with substance use in studies of adolescents and college students.
Change in self-reported impulsive behavior as measured by the 59-item Urgency, Premeditation, Perseverance, and Sensation Seeking Plus (UPPS-P) Impulsive Behavior scale (4 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  The Urgency, Premeditation, Perseverance, and Sensation Seeking Plus (UPPS-P) Impulsive Behavior scale is a 59-item self-report scale developed by Whiteside and Lynam to measure the multi-dimensional nature of impulsivity. Items are scored based on a four-point Likert-type scale as follows: 1) agree strongly, 2) agree somewhat, 3) disagree somewhat, and 4) disagree strongly. Factor analysis of eight other established scales that address impulsivity (in whole or part) revealed four factors that became the subscales in the UPPS-P: (lack of) Premeditation (11 items), Negative Urgency (11 items), Positive Urgency (14 items), Sensation Seeking (12 items), and (lack of) Perseverance (10 items). Internal consistency for these subscales showed alpha coefficients that ranged from 0.82 to 0.91.

SECONDARY OUTCOMES:
Change in self-reported soothability, planfulness, and distractibility as measured by the Kendall-Wilcox Self-Control Schedule (3 sub-scales). | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Soothability. The Soothability scale of the Kendall-Wilcox Self-Control Schedule assesses adolescents' capabilities to reduce emotional tension and control calmness when distressed. This 5-item scale includes items such as, "If I get annoyed about something, I can get over it pretty quick," and "I can easily calm down when I am excited or "wound up". Planfulness. This 7-item scale derived from the Kendall-Wilcox Self-Control Schedule assesses individuals' planfulness in everyday situations. Sample items include "I like to plan things way ahead of time." Distractibility. Adolescent tendency to be distracted from daily work is measured by a 6-item scale derived from the Kendall-Wilcox Self-Control Schedule. Sample items include "I like to switch from one thing to another."
Change in self-reported anger control and anger rumination as measured by the Children's Anger Management Scale (2 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Anger Control. Adolescents' anger management is assessed by the Anger Control subscale (4 items) of Children's Anger Management Scale (CAMS). Sample items include, "I can stop myself from losing my temper." Anger Rumination. The Anger Rumination subscale of the CAMS is used to measure an anger management domain of emotional SR. Items include, "I get angry thinking about things that happened in the past."
Change in self-reported sadness control and sadness rumination as measured by the Children's Sadness Management Scale (CSMS) (2 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Sadness Control. A 5-item subscale of the Children's Sadness Management Scale (CSMS) measures what adolescents might or might not do when they are feeling sad or down. The Sadness Control subscale includes items such as, "When I'm feeling down, I can control my sadness and carry on with things." Sadness Rumination. This 3-item measure for Sadness Rumination adapted from the CSMS assesses adolescents' emotional capabilities in dealing with sadness. Items include, "When people do something to make me sad, I don't forget about it."
Change in self-reported affective lability as measured by the Affective Lability Scale (originally 54 items, adapted to 10 items) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Affective Lability. A 10-item scale is adapted from the 54-item Affective Lability Scale. The Affective lability scale measures adolescents' tendency to change mood frequently. Sample items include, "My moods change a lot from day to day," and "I often switch back and forth from feeling irritated to feeling comfortable and relaxed."
Change in self-reported anger coping, problem solving, situation redefinition, impatience, and self-criticism as measured by the Wills Coping Inventory (5 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  The following subscales from the Wills Coping Inventory will be used: Anger coping, problem solving, situation redefinition, impatience, self-criticism.
Change in self-reported positive self-reinforcement as measured by the 8-item Heiby Self-Reinforcement Inventory | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Positive Self-Reinforcement. An 8-item scale is adapted from the Heiby Self-Reinforcement Inventory to measure adolescents' self-"reward" to prompt themselves to continue to perform a desired behavior. Items include "when I do something right, I take time to enjoy the feeling"
Change in self-reported present and future time perspective as measured by the Zimbardo Time Perspective Inventory (2 sub-scales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Future Time Perspective. An orientation toward present occurrences (e.g., seek out activities that produce immediate satisfaction such as alcohol use) versus future occurrences (e.g., invest in activities that require more effort but have positive long-term consequences such as physical exercise) has been considered to have significant effects on adolescent substance abuse: future orientation to have preventive effects and present orientation to have harmful effects on adolescent substance abuse and risky behaviors. This 7-item scale on Future Time Perspective is adapted from the Zimbardo Time Perspective Inventory (ZTPI). Items include "I am able to resist temptation when I know there is work to be done". Present Time Perspective. A 7-item scale on Present Time Perspective is derived from the ZTPI. Sample items include, "I think it's useless to plan too far ahead, because things hardly ever turn out the way I planned."
Change in self-reported impulsiveness as measured by the Eysenck Impulsiveness Questionnaire (EIQ) (1 subscale) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Impulsiveness. A 7-item scale from the Eysenck Impulsiveness Questionnaire (EIQ) assesses tendency for adolescents' impulsive responding. Sample items include "I often do things without stopping to think," and "I often get into trouble because I do things without thinking."
Change in self-reported substance use as measured by the Youth Risk Behavior Survey (YRBS) (4 subscales) | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Youth Risk Behavior Survey (YRBS) Middle School Version (http://www.cdc.gov/HealthyYouth/yrbs/index.htm). This is a nationally validated scale that measures substance use in children and adolescents. There are 16 questions in the substance use category of the 2013 middle school version of the YRBS for use of tobacco (8 questions), alcohol (2 questions), marijuana (2 questions), and other drugs (4 questions), taking approximately 10 minutes to complete. Each question includes an answer that allows participants to indicate whether they have ever used the substance, which will serve as a measure of use initiation over the time course of the entire study.
Change in self-reported substance use willingness as measured by the 13-item Substance Use Willingness Questionnaire | Baseline; 1 week post-intervention; 6 months post-intervention; 1 year post-intervention
  Substance Use Willingness Questionnaire. The Substance Use Willingness Questionnaire is composed of 13 items that ask how willing the participant would be to try cigarettes (3 questions), alcohol (3 questions), marijuana (3 questions), and other drugs (4 questions).

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir S Khalsa, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Boston Latin School, Boston, Massachusetts, United States